CLINICAL TRIAL: NCT02468518
Title: Randomized, Open Label Trial of Vitamin E on Change of Aerobic Bacterial Pattern
Brief Title: Effect of Vitamin E on Skin Aerobic Bacteria in Palmar Arsenical Keratosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Prof. Mir Misbahuddin, Prof. and Chairman, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BSMMU-007-CT
Record Dates: First submitted 2015-01-27; First posted 2015-06-11 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Arsenic Poisoning
MeSH Terms: interventions — Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patients (Experimental): Vitamin E capsule 200 IU bd x 12 weeks
  Interventions: Drug: Vitamin E capsule
- Arsenic exposed controls (Active Comparator): Vitamin E capsule 200 IU bd x 12 weeks
  Interventions: Drug: Vitamin E capsule
- Healthy volunteers (Active Comparator): Vitamin E capsule 200 IU bd x 12 weeks
  Interventions: Drug: Vitamin E capsule

INTERVENTIONS:
Drug: Vitamin E capsule — Capsules will be distributed to each participant free of cost
  Other Names: E-Cap, Batch No. 461016

SUMMARY:
This study will be conducted to observe any change in aerobic bacterial pattern on the skin of arsenicosis patients before and after administration of vitamin E (200 IU) capsules.

DETAILED DESCRIPTION:
Arsenicosis has emerged as one of the main and hazardous public health problem in Bangladesh. Melanosis and keratosis are the most common manifestations of arsenicosis. The exact mechanism of development of keratosis is not clear. With chronic ingestion of arsenic contaminated water the excretion of arsenic through skin increases and also the oxidative stress, which in turn cause cellular damage. These changes may influence the growth of normal bacteria and consistency of skin, which may be responsible for keratosis. In different study results shown that, vitamin E, a potential antioxidant that halts lipid peroxidation and maintains cell membrane integrity, also detoxified arsenic from the body. Normal skin bacteria mainly composed of Gram +ve bacteria. In arsenicosis, this pattern changes from Gram +ve bacteria to Gram -ve bacteria. Still now no study have been conducted to see, the effect of vitamin E on skin bacteria in arsenicosis, as skin bacteria changes. Therefore, this study will be conducted to observe any change in aerobic bacterial pattern on the skin of arsenicosis before and after administration of vitamin E capsules. Fifteen patients with skin manifestations, 15 arsenic exposed control, 15 healthy volunteers will be recruited on the basis of inclusion and exclusion criteria. They will be provide vitamin E capsules 200 IU twice daily for 12 weeks without any interruption. Water and nail samples will be collected for confirming the diagnosis. Skin samples will be collected two times (before and after giving vitamin E) for qualitative analysis of bacteria. All the patients, arsenic exposed controls and healthy subjects will be provided with same capsule in same dosage schedule. So, this study will find any change of skin bacteria pattern after administrating vitamin E capsule.

ELIGIBILITY:
Inclusion Criteria (Patients):

* History of drinking arsenic contaminated water (>50 µg/L) for more than 6 months
* Patients having moderate palmar keratosis
* Patients those voluntarily agree to participate

Inclusion Criteria (Arsenic exposed controls):

* Family members of the patient
* History of drinking arsenic contaminated water (>50 µg/L)
* Those voluntarily agree to participate
* No sign/symptoms of palmar keratosis

Inclusion Criteria (Healthy volunteers):

* Drinking arsenic safe water (<50 µg/L)
* Those voluntarily agree to participate

Exclusion Criteria:

* Pregnant and lactating mother
* Any other chronic disease like tuberculosis, diabetes, asthma
* Patients under treatment of arsenicosis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Identification of aerobic bacteria in five areas of the skin | 0 weeks (baseline), 12 weeks (end)
  Change in Number of aerobic bacteria in five areas (palm, dorsum of the hand, front of the chest, axilla and nare) of the skin of patients in comparison to arsenic exposed controls and healthy volunteers after 12 weeks of supplementation with vitamin E

SECONDARY OUTCOMES:
Clinical improvement in palmar arsenical keratosis following supplementation | 0 weeks (baseline), 12 weeks (end)
  There will be improvement of moderate palmar arsenical keratosis following supplementation with vitamin E

CONTACTS AND LOCATIONS:
Overall Officials: Mir Misbahuddin, Study Director — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Muradnagar Health Complex, Comilla, Bangladesh